CLINICAL TRIAL: NCT07261657
Title: A Pilot Trial of N-803 in Patients With Synovial Sarcoma and Myxoid/Round Cell Liposarcoma Previously Treated With Adoptive Cellular Therapy
Brief Title: N-803 in Patients With Progressive Synovial Sarcoma and Myxoid/Round Cell Liposarcoma Previously Treated With Adoptive Cellular Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 25S06; NCI-2025-08495 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00224911; NU 25S06 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Myxoid Liposarcoma; Round Cell Liposarcoma; Synovial Sarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma, Synovial | interventions — Specimen Handling; Leukapheresis; Magnetic Resonance Spectroscopy; ALT-803; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (N-803, leukapheresis) (Experimental): Patients receive N-803 SC on day 1 of each cycle. Cycles repeat every 14 days for up to 52 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo leukapheresis during screening up until day 1 cycle 1 and during treatment on day 8 cycle 4. Patients also undergo CT, chest x-ray, or MRI as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Biological: Nogapendekin Alfa Inbakicept; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nogapendekin Alfa Inbakicept — Given SC
  Other Names: ALT 803; ALT-803; ALT803; Anktiva; Fusion Protein Consisting of IL-15N72D and IL-15RASU/FC; IL-15N72D-IL-15RaSU/Fc; IL-15N72D/IL-15Ra-Fc; IL-15N72D:IL-15RaSu/Fc Fusion Complex; IL-15N72D:IL-15REC-SU/FC Soluble Complex I; Inbakicept Nogapendekin Alfa Fusion Complex; N 803; N-803; N803; Nogapendekin Alfa Inbakicept-pmln; Superagonist Interleukin-15:Interleukin-15 Receptor AlphaSu/Fc Fusion Complex Alt-803
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This early phase I trial tests the safety and how well N-803 works in treating patients with synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCL) that is growing, spreading, or getting worse (progressive) after being treated with adoptive cellular therapy (ACT) using T-cell receptor therapy (T-CRT). Synovial sarcoma is a rare, slow-growing cancer that affects the soft tissues, like muscles or ligaments near the joints. Myxoid/round cell liposarcoma is a rare type of soft tissue sarcoma cancer that originates from fat cells usually in the arms and legs. N-803 is a type of immunotherapy-a treatment that helps patients' own immune system fight cancer, and it is made up of a natural protein called interleukin-15 (IL-15) that is important for growing and activating immune cells. Studies have shown that patients can progress after initially responding to TCR-T, so this trial will use N-803 to stimulate rare persisting cells (cells that survive treatment and cause treatment failure and disease relapse) to make them work better at attacking the cancer. Adoptive cell therapy is a type of therapy that uses a patient's own immune cells to fight cancer. T-cell receptor therapy is a type of ACT that can recognize better recognize and bind to protein in cancer cells. Giving N-803 may be safe and tolerable in patients with SS or MRCL.

DETAILED DESCRIPTION:
CO-PRIMARY OBJECTIVES:

I. Assess whether nogapendekin alfa inbakicept (N-803) treatment in patients with SS and MRCL that received prior ACT using TCR-T cells expands rare persisting transferred TCR-T cells.

II. Assess the safety of N-803 in patients with SS and MRCL that received prior ACT using TCR-T cells.

SECONDARY OBJECTIVES:

I. Assess for preliminary evidence of N-803 clinical activity by imaging in patients with SS and MRCL that received prior ACT using TCR-T cells.

II. Evaluate 6-month progression free survival (PFS) of patients with SS and MRCL treated with N-803 and that have received prior ACT using TCR-T cells.

III. Evaluate median progression-free survival (PFS) of patients with SS and MRCL treated with N-803 and that received prior ACT using TCR-T cells.

EXPLORATORY OBJECTIVES:

I. To perform detailed phenotypic analysis of the persisting transferred T cells in pre-dose and on-treatment leukapheresis samples of patients with SS and MRCL treated with N-803 and that received prior ACT using TCR-T cells.

II. To perform detailed analysis of other immunologic subsets, including natural killer (NK) cells and monocytes, following patients with SS and MRCL treated with N-803 and that received prior ACT using TCR-T cells.

OUTLINE:

Patients receive N-803 subcutaneously (SC) on day 1 of each cycle. Cycles repeat every 14 days for up to 52 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo leukapheresis during screening up until day 1 cycle 1 and during treatment on day 8 cycle 4. Patients also undergo computed tomography (CT), chest x-ray, or magnetic resonance imaging (MRI) as well as blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed synovial sarcoma (SS) and/or myxoid/round cell liposarcoma (MRCL) who have progressed after ACT using TCR-T
* Patients must have been treated with a TCR-T product that can be assessed per medical history and/or discretion of the principal investigator. This includes the Food and Drug Administration (FDA) approved Afamitresgene autoleucel but also other products at the discretion of the principal investigator.

  * Note on references to Letetresgene Autoleucel and Afamitresgene Autoleucel: This study does not involve active treatment with TCR-T cell therapies, including Letetresgene autoleucel or Afamitresgene autoleucel. The investigational drug of this study is N-803
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Patients must have shown clinical benefit on at least one scan post ACT using TCR-T, (stable disease [SD], partial response [PR], complete response [CR]), as determined by the treating investigator
* Patients must be aged ≥ 18 to 80 at time of registration
* Patients must have a performance status of > 70% on the Karnofsky scale or < 2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Patients must be able to undergo leukapheresis per institutional standards. For patients receiving leukapheresis at the Rube Walker Blood Center, reference document guidance and Rube Walker Blood Center leukapheresis eligibility criteria
* Absolute lymphocyte count (ALC) ≥ Institutional lower limit of normal (within screening window of 28 days up until pre-dose leukapheresis)
* Absolute neutrophil count (ANC) ≥ 1,000/mcL (within screening window of 28 days up until pre-dose leukapheresis)

  * Prior growth factors are allowed per treating investigator discretion (i.e. erythropoietin [EPO]), granulocyte-macrophage colony-stimulating factors (GM-CSF) such as sargramostim, platelet-derived growth factor (PDGF), granulocyte colony-stimulating factors (G-CSF) including filgrastim, darbepoetin alfa are allowed per standard of care
* Hemoglobin (Hgb) ≥ 8.3 g/dL (within screening window of 28 days up until pre-dose leukapheresis)
* Platelets (PLT) ≥ 40,000/mcL (within screening window of 28 days up until pre-dose leukapheresis)
* Total bilirubin ≤ Institutional upper limit of normal (ULN) (within screening window of 28 days up until pre-dose leukapheresis)

  * Unless the patient has documented Gilbert's syndrome. Patients with Gilbert syndrome may be eligible with total bilirubin up to 3 × ULN, provided direct bilirubin is within normal limits and per investigator discretion
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 1.5 x institutional ULN (within screening window of 28 days up until pre-dose leukapheresis)
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 1.5 x institutional ULN (within screening window of 28 days up until pre-dose leukapheresis)
* Alkaline phosphatase (ALP) ≤ 2.5 institutional ULN (within screening window of 28 days up until pre-dose leukapheresis)
* Serum creatinine ≤ 2.0 mg/dL or 177 μmol/L or creatinine clearance ≥ 40 mL/min (using the Cockcroft-Gault formula) (within screening window of 28 days up until pre-dose leukapheresis)
* Note: All laboratory value permitted departures (described in the above table with a different ULN) should be clearly documented by the treating investigator in the sources
* Note: Patients do not need to meet lab eligibility requirements after screening. For days of leukapheresis, refer to institutional guidelines for lab eligibility for leukaphereses (see Rube Walker Blood Center leukapheresis eligibility criteria)
* Note: The institutional upper limit refers to the reference range upper limit established by the institution where the laboratory tests were performed
* The effects of N-803 on the unborn fetus are unknown. For this reason, patients of child-bearing potential (POCBP) and their partners with sperm-producing reproductive capacity must agree to use adequate contraception from start of treatment, for the duration of study participation, and for 7 months following completion of N-803 therapy. Should a POCBP become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. Patients with sperm-producing reproductive capacity (PWSPRC) treated or enrolled on this protocol must also agree to use adequate contraception with partners of childbearing potential from time of informed consent, for the duration of study participation, and 7 months after completion of administration

  * Note: A POCBP is any patient (regardless of gender, sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) with an egg-producing reproductive tract who meets the following criteria

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative pregnancy test during screening and per the study schedule. See study procedures for more information
* Patients must have the ability to understand and the willingness to sign a written informed consent document and comply with the study requirements

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, neuropathy and other non-significant adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v 5.0) as deemed by the principal investigator
* Any medical diagnosis that would prevent the donation of white blood cells (WBCs) or patients whom in the opinion of the investigator should not donate WBCs
* Patients with high risk of bleeding, as determined by treating investigator.

  * Note: If patients are on anticoagulants, the investigator will determine if patient can continue anticoagulants throughout the study, or if their dosage needs to be changed until completion of both leukapheresis procedures
* Patients with illnesses or conditions that would prevent them from taking blood thinners or patients whom in the opinion of the investigator should not take blood thinners
* Patients who have received other IL-15 treatments since receiving TCR-T cells to the start of study treatment (C1D1).

  * Note: Prior growth factors are allowed per treating investigator discretion (i.e. erythropoietin (EPO), granulocyte-macrophage colony-stimulating factors (GM-CSF) such as sargramostim, platelet-derived growth factor (PDGF), granulocyte colony-stimulating factors (G-CSF) including filgrastim, darbepoetin alfa
* Patients with new or progressing brain metastases.

  * Note: Patients with treated brain metastases that are stable in the opinion of the treating investigator are eligible
* Known significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to pre-dose leukapheresis, unstable arrhythmias, or unstable angina. To be eligible for this trial, patients should be class 2B or better
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to N-803 or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Participants who, in the opinion of the investigator, are unable to safely or feasibly receive subcutaneous injections of N-803. Examples include:

  * Absence of suitable subcutaneous tissue for injection (e.g., due to cachexia, scarring, or anatomical limitations).
  * Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to N-803, or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
  * Active skin conditions or infections at potential injection sites.
  * Physical or psychological inability to tolerate subcutaneous injection procedures (e.g., severe needle phobia, movement disorders).
  * Medical contraindications to subcutaneous administration (e.g., bleeding disorders, severe dermatologic conditions).
  * Any other factors that, in the judgment of the investigator, would interfere with safe and feasible administration of subcutaneous injections
* Major surgical procedure (e.g., gastrointestinal [GI] surgery, removal or biopsy of brain metastasis), other than for diagnosis or known need for a major surgical procedure while on study treatment.

  * Note: Patients must have fully recovered from complete wound healing from said surgery prior to first study assessment, in the opinion of the treating investigator.
  * Note: Surgery and radiation are allowed after completion of cycle 5 per discretion of treating investigator (CT scan and N-803 administration at cycle 5 must have already occurred)
* Systemic autoimmune disease currently requiring treatment (e.g., lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma). The patient must have been off treatment for 90 days from registration
* History of organ transplant requiring immunosuppression; or history of pneumonitis or interstitial lung disease requiring treatment with systemic steroids; or a history of receiving systemic steroid therapy or any other immunosuppressive medication ≤ 3 days prior to study initiation. Daily steroid replacement therapy (e.g., prednisone or hydrocortisone at doses of ≤ 10 mg/day of prednisone (or equivalent)) and corticosteroids used to manage adverse events (AEs) are permitted. Patients who require immunosuppressive agents during their study participation are ineligible, except:

  * Use of physiologic doses of systemic steroid replacement is permitted at doses of ≤ 10 mg/day of prednisone (or equivalent, e.g., dexamethasone 1.5 mg, methylprednisolone 8 mg, or hydrocortisone 40 mg).
  * Local steroids, including topical steroids (e.g., hydrocortisone, clobetasol), nasal steroids (e.g., fluticasone, mometasone), or inhaled steroids (e.g., budesonide, beclomethasone).
  * Limited courses (< 1 week) of systemic steroids (≤ 10 mg/day of prednisone or equivalent) (e.g, in patients with exacerbations of reactive airway disease or anaphylaxis in patients who have known contrast allergies).
  * Immunosuppressive treatments to optimally manage immune-related AEs as clinically indicated
* Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the patient at high risk for treatment-related complications
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment including:

    * Known active infection with acute or chronic hepatitis B or C, known active human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome
    * Exception: uncomplicated urinary tract infections (or sinus infections and are on antibiotics)
  * (AIDS)-related illness
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen except the following:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * In situ cervical cancer that has undergone potentially curative therapy
* Patient is pregnant or nursing.

  * Note: Pregnant patients are excluded from this study because N-803 is an interleukin-15 (IL-15) receptor agonist with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with N-803, breastfeeding should be discontinued if the mother is treated with N-803
  * Note: Serum test will be conducted at screening (serum pregnancy test [beta-human chorionic gonadotropin [β-HCG])
* Other conditions which, in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study
* Patients who need to be on concurrent anticancer treatment (e.g., chemotherapy, immunotherapy, cytokine therapy [except erythropoietin]) throughout participation in the study
* Patients who have had prior use of narrow therapeutic index drugs that are substrates of major CYP450 enzymes within 28 days of first study drug administration per discretion of the treating investigator, including but not limited to:

  * Tacrolimus
  * Cyclosporine
  * Sirolimus
  * Everolimus
  * Warfarin
  * Phenytoin
  * Midazolam
  * Tamoxifen
  * Codeine
  * Erlotinib
* Patients who have had prior use concomitant medications that prolong the QT/corrected QT (QTc) interval within 28 days of first study drug administration visit per discretion of the treating investigator
* Patients who have had prior biologic therapies or chemotherapy within 28 days of pre-dose leukapheresis visit, or radiation therapy within 14 days of pre-dose leukapheresis visit
* Patient must have reviewed and signed the informed consent document before any study activities may occur. Registration of patients is completed in NOTIS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-09-02 (Estimated); Primary Completion 2030-09-02 (Estimated); Study Completion 2032-09-02 (Estimated)

PRIMARY OUTCOMES:
The expansion of rare persisting transferred T-cell receptor therapy | Before and after eight weeks of N-803 therapy
  Will be assessed using T-cell receptor sequencing or flow cytometry.
Incidence of adverse events | Up to 30 days after the last administration of N-803
  Will be determined by the incidence, severity, and attribution of adverse events graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Overall response rate | Up to 4 years
  Will be defined by Response Evaluation Criteria in Solid Tumors version 1.1. Will be estimated with a two-sided 95% confidence interval using the Clopper-Pearson method.
Six-month progression-free survival (PFS) | Up to 4 years
  Defined as the proportion of patients who remain alive and progression-free at six months (± 2 weeks) from treatment initiation. The Kaplan-Meier method will be used to estimate the six-month PFS rate, and a corresponding 95% confidence interval will be reported.
Median PFS | Up to 4 years
  Kaplan-Meier curves will be reported descriptively, and median PFS will only be interpreted if the survival function drops below 50% with sufficient events to support stable estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Seth M Pollack, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States